CLINICAL TRIAL: NCT04901507
Title: Effects of an External Oral Irrigation Device on Patients With Dry Mouth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Voutia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM20021188
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- The Voutia System (Experimental): The Voutia System oral irrigation device
  Interventions: Device: The Voutia System

INTERVENTIONS:
Device: The Voutia System — Participants will wear the Voutia System oral irrigation device continuously through the day and night, removing for cleaning and if otherwise necessary, but not for time extending beyond six-eight hours.
  Other Names: Oral irrigation device

SUMMARY:
The purpose of this research study is to test the effectiveness of treating dry mouth through water rehydration using this extra oral water pump/irrigation device.

DETAILED DESCRIPTION:
Dry mouth causes difficulty with chewing, swallowing, speech, and increases the risk dental cavities. It also can cause discomfort in the mouth, and a loss of general quality of life. The oral irrigation device supplies a small amount of water to participant's mouth through a small tube that is placed in the corner of the mouth throughout the time participants wear it.

In this study, participants will be asked to:

1. Visit the dental school clinic two (2) times for study visits.
2. Wear the oral irrigation device as directed by the investigator.
3. Keep notes at home.
4. Answer survey questions during both dental visits about dry mouth symptoms.
5. Give permission for the researchers to collect information about medications or health conditions that contribute to dry mouth from participant's medical records.

ELIGIBILITY:
Inclusion Criteria:

* patients who report xerostomia (dry mouth) and are diagnosed after testing with hypofunctioning salivary glands

Exclusion Criteria:

* Patient who after testing do not exhibit salivary hypofunction
* Children
* Patient with limited English proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susie Goolsby, DDS, MSHA, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Voutia System
Started | 16
Completed | 13
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | The Voutia System
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1
  Race: Black/African American | 2
  Race: White/Caucasian | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16
CODS [Mean (Standard Deviation); unit: units on a scale] — Clinical Oral Dryness Score- a clinician scored features observed in the patient's mouth and derived a COD score of 0-10. Clinical findings observed were given a one-point value towards the CODS, with 10 indicating the most severe oral dryness. Population: Three subjects withdrew prior to baseline outcome measures being recorded. Three subjects withdrew prior to baseline outcome measures being recorded.
  units on a scale
    number analyzed (Participants) | 13
    (all) | 6.6 (2.2)
OHIP [Mean (Standard Deviation); unit: units on a scale] — Oral Health Impact Profile (OHIP-14) used to measure Oral Health-Related Quality of Life (OHRQoL) Population: Three subjects withdrew prior to baseline outcome measures being recorded.
  units on a scale
    number analyzed (Participants) | 13
    (all) | 33.1 (14.05)
Xerostomia Inventory [Mean (Standard Deviation); unit: units on a scale] — Population: Three subjects withdrew prior to baseline outcome measures being recorded.
  units on a scale
    number analyzed (Participants) | 13
    (all) | 46.4 (9.06)

OUTCOME MEASURES:

1. Primary Outcome: Change in Oral Health Related Quality of Life (OHRQoL)
Description: OHRQoL will be assess using the Oral Health Impact Profile (OHIP-14). The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items on the scale. Higher OHIP-14 scores indicate worse and lower scores indicate better OHRQol
Time Frame: Baseline to 4 - 6 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | The Voutia System
Number analyzed (Participants) | 13
score on a scale | 10.2 [0.07 to 20.24]

2. Primary Outcome: Change in Oral Health Related Quality of Life - Dry Mouth Specific (OHRQoL-XI)
Description: OHRQoL-XI will be assessed using the Xerostomia Inventory (XI), an 11-item summated rating scale which combines the responses to 11 individual items into a single continuous scale score which represents the severity of chronic xerostomia. Scores range from 11 to 55 with higher scores represent more severe symptoms.
Time Frame: Baseline to 4 - 6 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | The Voutia System
Number analyzed (Participants) | 13
score on a scale | 13.2 [6.0 to 20.4]

3. Primary Outcome: Change in Oral Dryness
Description: Clinical Oral Dryness Score (CODS) conducted during the clinical exam assesses ten key features of dry mouth and allocates one point for each feature. The total score ranges from 0 to 10 with higher scores indicating more severe dry mouth.
Time Frame: Baseline to 4 - 6 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | The Voutia System
Number analyzed (Participants) | 13
score on a scale | 0.85 [-0.04 to 1.73]

4. Primary Outcome: Clinical Changes in Stimulated Saliva Flow
Description: Data on routine stimulated saliva testing as performed as standard of care for patients suspected to have reduced salivary flow will be compared before and after use of the device.
Time Frame: Baseline to 4 - 6 weeks
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | The Voutia System
Number analyzed (Participants) | 13
mL/min | 0.73 [0.11 to 1.36]

5. Primary Outcome: Clinical Changes in Unstimulated Saliva Flow
Description: Data on routine unstimulated saliva testing as performed as standard of care for patients suspected to have reduced salivary flow will be compared before and after use of the device.
Time Frame: Baseline to 4 - 6 weeks
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | The Voutia System
Number analyzed (Participants) | 13
mL/min | 5.7 [-1.6 to 12.9]

ADVERSE EVENTS:
Time Frame: Study subjects utilized the Voutia device for a period of approximately 2 months during which time adverse events were monitored.
Arm/Group | The Voutia System
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04901507/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04901507/SAP_003.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT04901507/ICF_002.pdf